CLINICAL TRIAL: NCT04204707
Title: PROCURE: Patient Reported Outcomes After Surgery for Deep Endometriosis Infiltrating the Muscular Layer of the Rectum: a Prospective Study
Brief Title: Patient Reported Outcomes After Surgery for Rectal Endometriosis
Acronym: PROCURE
Status: Active, not recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Semmelweis University (Other)
Responsible Party: Sponsor
Other Study IDs: S62986
Record Dates: First submitted 2019-12-16; First posted 2019-12-19 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Endometriosis; Endometriosis, Rectum; Endometriosis-related Pain; Endometriosis; Bowel
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Conservative surgery
  Interventions: Other: PROMS
- Radical surgery (segmental resection)
  Interventions: Other: PROMS

INTERVENTIONS:
Other: PROMS — Patient Reported Outcomes after different types of surgery for rectal endometriosis

SUMMARY:
To describe the difference in patient reported outcomes after conservative treatment in comparison to radical rectal surgery in patients with deep endometriosis infiltrating the rectum (up to 15cm from the anus with at least involvement of the muscularis layer) and to determine predictors for radical surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 - 45 years (both inclusive)
* BMI <35
* Complaining of infertility and/or pain
* Deep endometriosis infiltrating the rectum on at least one imaging technique up to 15 cm from the anus and involving at least the muscularis layer in depth

Exclusion Criteria:

* Refusal of bowel resection/stoma
* History of laparotomy for endometriosis
* (history of) Hysterectomy
* Suspected pelvic malignancy
* Pregnancy
* Impossibility for postoperative follow-up in our hospital

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: Women scheduled for a multidisciplinary laparoscopic surgery for rectal endometriosis.
Sampling Method: Probability Sample
Enrollment: 294 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients experiencing one of the following symptoms at 12 months postoperatively: | 12 months postoperatively
  * constipation (1 stool/>5 consecutive days)
  * frequent bowel movement (≥3 stools/day)
  * defecation pain
  * anal incontinence (involuntary loss of gas or stools)
  * dysuria
  * bladder atony requiring self-catheterization
The determination of possible risk factors for radical surgery. | 3 months postoperatively
  based on patient complaints, preoperative imaging techniques and intra operative finding

CONTACTS AND LOCATIONS:
Overall Officials: Carla Tomassetti, MD, PhD, Principal Investigator — UZ Leuven
Locations (2):
- UZ Leuven, Leuven, Belgium
- Semmelweis University Hospital, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No